CLINICAL TRIAL: NCT01536756
Title: A Single Blind Randomized Controlled Study Investigating the Effectiveness of a Structured Physical Rehabilitation Program on the Physical Fitness and Negative Psychological Symptoms for Chinese Patients With Mild to Severe Depressive Disorders
Brief Title: Effectiveness of a Structured Physical Rehabilitation Program for Chinese Patients With Depressive Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kowloon Hospital, Hong Kong (Other)
Collaborators: Kwai Chung Hospital (Other)
Responsible Party: Principal Investigator, Dr. Lau Mo Yee Polly, Cluster Manager (Physiotherapy), Kowloon Central Cluster, Kowloon Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KH-KCH-PSY-RCT
Record Dates: First submitted 2012-02-10; First posted 2012-02-22 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Depressive Disorders
Keywords: Depressive disorder; exercise; pain; physical; psychological; Chinese; mild to severe depressive disorders
MeSH Terms: conditions — Depressive Disorder; Motor Activity; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Intervention -- Physical Rehabilitation Program (Experimental)
  Interventions: Other: Exercise Intervention -- Physical Rehabilitation Program
- Wait List Control Group (Other)
  Interventions: Other: Wait List Control Group

INTERVENTIONS:
Other: Exercise Intervention -- Physical Rehabilitation Program — The intervention group will participate in a "Physical Rehabilitation Program" which includes a 60-minute training session at a frequency of 3 times a week over a total of 12-week duration. The training session consists of 45 minutes of warm-up stretching and circuit training. This includes 3 stations of aerobic exercises for physical work up of different body parts, and 3 stations of strengthening exercises of major muscles groups at 3 sets of 10 repetitions. The final 15-minute training session will be the cooling down exercise with emphasis on stress management incorporating mindful breathing, stretching and body awareness exercise.
  Arms: Exercise Intervention -- Physical Rehabilitation Program
Other: Wait List Control Group — The subjects of the control group will be asked to maintain their usual activities while awaiting for the physical rehabilitation program at the 12-week waiting time. They will be allowed to receive any other usual medical services including social services and psychotherapy but not physiotherapy services. At the end of the 3rd month, the control group will be recruited into the Physical Rehabilitation Program. Patients in the control group will then join in as the intervention group and follow the intervention and assessment protocol.
  Arms: Wait List Control Group

SUMMARY:
Evidence shows that depression was found to be associated with physical inactivity and on the other hand, high prevalence of depression was also found in patients with chronic pain. Structured physical rehabilitation program with exercises as main component and pain management provided by physiotherapy has been proved by overseas studies to be effective in reducing the psychological symptoms of depression through increasing the physical fitness and relieving the pain. Literatures also reported a strong sociocultural influence on the prevalence of depression and the manifestations of their clinical signs and symptoms in patients suffered from mental health problems between Chinese and Western societies. The benefits of physical rehabilitation program in the management of depression cannot be assumed in the Chinese population. The purpose of this study is to investigate the effectiveness of a structured "Physical Rehabilitation Program" for Chinese patients diagnosed with depressive disorder (mild to severe severity) on the physical fitness and negative psychological symptoms of the recruited patients.

The Hypothesis are:

1. The Physical Rehabilitation Program is effective in improving the physical fitness in Chinese patients with depressive disorders.
2. The Physical Rehabilitation Program is effective in alleviating the negative psychological symptoms in Chinese patients with depressive disorders.

DETAILED DESCRIPTION:
Eighty-four Chinese patients who are diagnosed as depressive disorders with age between 18 and 64 years old, fulfilling the inclusion criteria (stated at the attached study proposal) will be recruited for a 12-week physical rehabilitation program with forty-two patients for the intervention group (n=42) and equal sample size for the control group (patient put on the waiting list for the Physical Rehabilitation Program). All patients will be allocated to either the intervention group or control group by computer generated block randomization with block size of 6 persons using StatsDirect Software, version 2.7.8. The subjects of the control group will be asked to maintain their usual activities while awaiting for the physical rehabilitation program at the 12-week waiting time. They will be allowed to receive any other usual medical services including social services and psychotherapy but not physiotherapy services. At the end of the 3rd month, the control group will be recruited into the Physical Rehabilitation Program. Patients in the control group will then join in as the intervention group and follow the intervention and assessment protocol. All the patients will be instructed not to disclose their grouping to the assessor. Sub-group analysis will be conducted for further in-depth analysis of the subjects in the intervention group having clinical manifestations of pain interference as triage by the 7 items in Brief Pain Inventory (BPI) - short form - Chinese version. Outcome measures on the physical and mental domains will be conducted: at baseline (T1-before commencement of program), end of the 3rd month (T2-end of program for intervention group; end of the waiting time of control group), 12 months (T3-one year long term follow-up for the intervention group). Validity and reliability of all the adopted outcome measures were reported in medical literatures. There is no reported harmful effect on all interventions and there is no pain or discomfort for all of the testing procedures. Physical outcome measures include body composition (body mass index, percentage of body fat); flexibility (sit and reach flexibility); muscular endurance (1-minute sit-up count); muscle strength (hand grip strength, isometric quadriceps strength); cardiovascular endurance (maximal oxygen consumption) and physical functioning (Brief Pain Inventory- Chinese version). Mental outcome measures include depression, anxiety & stress (Depression, Anxiety, Stress Scale (DASS-21) - Chinese version); depression (Hamilton Depression Rating Scale- Chinese version) and self-esteem (Rosenberg Self-Esteem Scale- Chinese version). The findings will serve as pilot program for rolling out of the services for Chinese patients with depressive disorders to other clusters / hospital and reference base for future territory-wide profile study on this clientele and randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18 and 64 Chinese adults with diagnosed depressive disorders of mild to severe severity (Diagnostic code: F32.0 to F33.9 under International Classification of Diseases, 10th revision) as referred from the Department of Psychiatry of Kowloon Hospital or Kwai Chung Hospital;
2. Able to read, write and understand Chinese;
3. Mentally capable of making written consent for participation of the study.

Exclusion Criteria:

1. Unstable medical and/or psychological states such as suicidal risk and aggressive impulses, or severe cognitive, language, or hearing deficits;
2. Orthopaedic problems or other diseases which limit physical fitness assessment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Body Composition at 3 months and 12 months | Baseline, 3 months and 12 months
  Body Mass Index & Percentage of Body Fat
Change from Baseline in Flexibility at 3 months and 12 months | Baseline, 3 months and 12 months
  Sit and Reach Flexibility
Change from Baseline in Muscle Strength at 3 months and 12 months | Baseline, 3 months and 12 months
  Hand Grip Strength & Quadriceps Strength
Change from Baseline in Muscular Endurance at 3 months and 12 months | Baseline, 3 months and 12 months
  One-Minute Sit-up Count
Change from Baseline in Cardiovascular Endurance at 3 months and 12 months | Baseline, 3 months and 12 months
  Maximal Oxygen Consumption
Change from Baseline in Physical Functioning at 3 months and 12 months | Baseline, 3 months and 12 months
  pain interference score of Brief Pain Inventory- Chinese version

SECONDARY OUTCOMES:
Change from Baseline in Depression, Anxiety and Stress at 3 months and 12 months | Baseline, 3 months and 12 months
  Depression Anxiety Stress Scale - 21 - Chinese Version
Change from Baseline in Depression at 3 months and 12 months | Baseline, 3 months and 12 months
  Hamilton Depression Rating Scale- Chinese version
Change from Baseline in Self-esteem at 3 months and 12 months | Baseline, 3 months and 12 months
  Rosenberg Self-Esteem Scale- Chinese version

CONTACTS AND LOCATIONS:
Overall Officials: Mo Yee P Lau, DHSc, Principal Investigator — Kowloon Hospital, Hong Kong
Locations (2):
- China (2):
  - Physiotherapy Department, Kowloon Hospital, Hong Kong
  - Physiotherapy Department, Kwai Chung Hospital, Hong Kong

REFERENCES:
- [Derived] Chau RMW, Tsui AYY, Wong EYW, Cheung EYY, Chan DYC, Lau PMY, Ng RMK. Effectiveness of a structured physical rehabilitation program on the physical fitness, mental health and pain for Chinese patients with major depressive disorders in Hong Kong - a randomized controlled trial with 9-month follow-up outcomes. Disabil Rehabil. 2022 Apr;44(8):1294-1304. doi: 10.1080/09638288.2020.1800833. Epub 2020 Aug 8. PMID 32772583